CLINICAL TRIAL: NCT03139201
Title: A Prospective Randomized Controlled Study to Evaluate the Clinical Performance of OxyAqua Silicone Hydrogel Soft Contact Lens
Brief Title: Clinical Performance of the OxyAqua Daily Disposable Silicone Hydrogel Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visco Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1040625M
Record Dates: First submitted 2017-04-29; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Myopia
Keywords: silicone hydrogel soft contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OxyAqua (Experimental): OxyAqua (olifilcon D) daily disposable
  Interventions: Device: OxyAqua
- Si-Hy (Active Comparator): Si-Hy (olifilcon B) daily disposable
  Interventions: Device: Si-Hy

INTERVENTIONS:
Device: OxyAqua — OxyAqua (olifilcon D) silicone hydrogel soft contact lens
  Arms: OxyAqua
Device: Si-Hy — Si-Hy (oliflcon B) silicone hydrogel soft contact lens
  Arms: Si-Hy

SUMMARY:
The objective of this study is to demonstrate that the OxyAqua silicone hydrogel soft contact lens could be prescribed as a supportive care for myopes.

DETAILED DESCRIPTION:
This is a double blind randomized control study to evaluate a daily disposable contact lens. It is planned to have 30 evaluable subjects at least divided evenly among 3 independent PIs from one hospital. Each PI will enroll 12 subjects at least. The ration of evaluable test subjects to control subjects will be 2 to 1. The study lens will be dispensed randomly to subjects who have normal ocular health and conform to a set of criteria. It is necessary to wear the lens 8 hours a day and 5 days a week at least and follow up for one month (30 days). Data will be collected at baseline, 1 week, 2 week and 4 week of daily disposable modality including Adverse Reactions, Slit-lamp findings and Symptoms, Problems, and Complaints, vision acuity, keratometry change and reason for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have normal eyes and use no ocular medications. They may have worn contact lenses previously, provided their eyes are shown to be normal at the start of the investigation. A normal eye is defined as having the following characteristics:

  1. No anterior segment infection, inflammation or abnormality.
  2. No other active ocular or systemic disease that would contraindicate contact lens wear; and
  3. No medications that would contraindicate contact lens wear.
* VA correctable to 0.1 LogMAR or better, with spherical lenses ranging in power from
* 1.00 to -10.00 D myopia, astigmatism less than 2.00 D
* Willing to comply with all study procedures and be available for the duration of the study.
* Provide signed and dated informed consent form.

Exclusion Criteria:

* Have history of allergies that would contraindicate "normal" contact lens wear.
* Have other active ocular or systemic disease such as, but not limited to: anterior uveitis (past or present), glaucoma, Sjögren's syndrome, lupus erythematosus, sclerodermas, keratoconus or type II diabetes, slip lamp findings greater than grade I (such as cornea or interstitial edema).
* Have medications that would contraindicate contact lens wear.
* Have had any cornea surgery.
* Currently pregnant (to the best of the subject's knowledge), is lactating or is planning a pregnancy within the next 1 month.
* Any active participation in another clinical trial within 30 days prior to this study.
* The presence of clinically significant (grade 3 or 4) anterior segment abnormalities; inflammations such as iritis; or any infection of the eye, lids, or associated structures.
* A known history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates or fungal infections.
* A history of papillary conjunctivitis that has interfered with contact lens wear.
* No monocular or monovision fits.
* Alcoholic or Drug Abused.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2016-12-08 (Actual); Study Completion 2016-12-08 (Actual)

PRIMARY OUTCOMES:
Log MAR visual acuity (VA) | one month
  the visual acuity corrected with contact lens could reach 0.1 or better

SECONDARY OUTCOMES:
Any slit lamp findings > grade 2 | over all follow-up visits for the 1 month
  slit lamp findings on all dispensed eyes over all follow-up visits. Measured on a scale of 0-4 with 0=no findings and 4=sever findings.
Subjective response to comfort, symptoms and complaints | over all follow-up visits for the 1 month
  subjective ratings of comfort, symptom and complaints using a scale of 0=severe stinging/Burning to 5=No stinging/Burning for each eye

CONTACTS AND LOCATIONS:
Overall Officials: Huey Chuan Cheng, MD MDS, Study Director — Mackay Memorial Hospital; Shu-I Yeh, MD MS, Principal Investigator — MacKay Memorial Hospital - Tamshui; Jy Been Liang, MD, Principal Investigator — Tri-Service General Hopsital - Tingjhou Branch

IPD SHARING:
Plan to Share IPD: No